CLINICAL TRIAL: NCT04656171
Title: Microcephaly, Fanconi Anemia and Praxial Disorders
Acronym: MicroFancII
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No financement AFAM
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP200090; N° IDRCB: 2019-A03171-56 (Registry Identifier: ANSM)
Record Dates: First submitted 2020-11-05; First posted 2020-12-07 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Fanconi Anemia
MeSH Terms: conditions — Fanconi Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minor patients with Fanconi anemia (Experimental): MRI of hands and forearm, neuropsychological and neuromotor tests
  Interventions: Radiation: MRI of the hand and forearm,
- Minor controls (Active Comparator): MRI of the hand and forearm, orthopedic evaluation, neuromotor tests of the upper limbs, praxies evaluation, neurocognitive evaluation
  Interventions: Radiation: MRI of the hand and forearm,

INTERVENTIONS:
Radiation: MRI of the hand and forearm, — MRI of the hand and forearm,

SUMMARY:
Fanconi Anemia (FA) is mentioned in children with congenital malformations including kidney, hart and skeletal malformations (absence or abnormal thumb or forearm), and bone marrow failure or myelodysplasia with a progressive onset in childhood or adulthood. No study has focused on microcephaly, a reduction in brain volume, which is present in 20% of children, and its consequences on cognitive and structural level of the brain. Since 2014, Robert-Debré's team has been interested in this functional cognitive and neuroanatomical approach trough a National PHRC. Preliminary results carried out on 12 children show that their intellectual efficiency was in the normal range for age. However, we noticed a significant difference between abilities in comprehension and verbal reasoning corresponding to what is expected for age, and the sensorimotor skills or fine motor praxia significantly reduced. These difficulties, graphically penalizing for these children, are not always explained by a skeletal malformation of the upper limb, suggesting that musculo-tendinous anomalies may be associated. The objectives of our project are: 1) to identify upper limb musculo-tendinous abnormalities and their functional consequences, 2) to determine if these abnormalities could influence the somatosensory representation of the upper limb at the cerebral cortical level. This project should help us to better understand the fine motor disabilities or developmental coordination disorder of these children, which penalize their learning, and provide them with adapted solutions.

DETAILED DESCRIPTION:
Our hypothesis is that children with FA present a developmental dyspraxia. This condition is very penalizing for children especially regarding graphic tasks, handwriting, whether or not they have skeletal malformations of the upper limbs. Consequences are fatigue because of energy expended trying to execute fine motor movements correctly.

Main objective:

To identify gesture dyspraxia in order to propose a targeted rehabilitation leading to national recommendations.

Main Evaluation Criteria :

1. measurement of fine motor praxia
2. quantification of dyspraxia

Secondary Objectives :

To identify the musculoskeletal or tendinous anomalies in the upper limbs of AF children and to assess their functional consequences.

To determine if these upper limbs abnormalities could influence the somatosensory map of this part of the body in the cerebral cortex.

Secondary Evaluation Criteria :

1. MRI of the hand and forearm, orthopedic examination and functional assessment
2. Previously obtained brain MRI data

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Fanconi Anemia defined according to two of the following diagnostic criteria already included in the MicroFanc study:

   * Chromosome breakage test after exposure to an alkylating agent (mitomycin) on peripheral blood lymphocytes.
   * FancD2 test on lymphocytes or fibroblasts
   * sensitivity of fibroblasts to mitomycin
   * mutation in one of the FANC complementation genes (A, B, C, D1, D2, E, F, G, I, J, L, M, N)
2. Non-transplanted patients or patients at a distance from CSH transplant (>3 years)
3. Age ≥5 years of age at inclusion (minimum age of accessibility for neuropsychological tests and no need for sedation for MRI)

Exclusion Criteria:

Subjects for whom both parents have not agreed to participate in the research, or for whom MRI is contraindicated.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
measurement of fine motor praxia | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Passemard, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Drbré Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No